CLINICAL TRIAL: NCT05731999
Title: A First-in-human Explorative Pilot Study in Healthy Volunteers Measuring Eye Parameters With a New Mobile Phone Application for Future Monitoring of Patients in Treatment of Substance Use Disorder
Brief Title: A First Study in Healthy Volunteers of a New Mobile Phone Application Measuring the Eyes Before and After Medication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kontigo Care AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KCClin01
Record Dates: First submitted 2023-01-30; First posted 2023-02-16 (Actual); Results first posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Drug Abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to one out of four arms, i.e., single application of either phenethylamines, benzodiazepines, cannabinoids, or opioids. The investigation aims to enroll 11 subjects, i.e., healthy volunteers, per medicinal product group that have completed the clinical investigation until the telephone follow-up call. For four medicinal products, the total will be 44 subjects. In order to take account for a drop-out rate of 10%, 12 subjects will be included per medicinal product group and in total 48 subjects in the clinical investigation. As this is an early feasibility and explorative investigation, the sample size is not derived from a sample size calculation as no hypothesis is pre-defined.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Single application of phenethylamines (D1) (Experimental): Evaluation of Previct Drugs' function to measure pupils and eye movements and to evaluate if there are any changes in the pupillometric parameters before and after intake of phenethylamines.
  Interventions: Device: Previct Drugs
- Single application of benzodiazepines (D2) (Experimental): Evaluation of Previct Drugs' function to measure pupils and eye movements and to evaluate if there are any changes in the pupillometric parameters before and after intake of benzodiazepines.
  Interventions: Device: Previct Drugs
- Single application of cannabinoids (D3) (Experimental): Evaluation of Previct Drugs' function to measure pupils and eye movements and to evaluate if there are any changes in the pupillometric parameters before and after intake of cannabinoids.
  Interventions: Device: Previct Drugs
- Single application of opioids (D4) (Experimental): Evaluation of Previct Drugs' function to measure pupils and eye movements and to evaluate if there are any changes in the pupillometric parameters before and after intake of opioids.
  Interventions: Device: Previct Drugs

INTERVENTIONS:
Device: Previct Drugs — Previct Drugs is a new non CE-marked eHealth system intended to be used for future monitoring and treatment of patients with substance use disorder (SUD). Previct Drugs consists of an application (app) to be installed on a smartphone, a web-based careportal to be accessed from a computer by the healthcare professional for administration and access of registered data, and a database for storage, handling, and analysis of reported data. Previct Drugs is intended to be used by healthcare professionals and patients within treatment of SUD.

SUMMARY:
This is a pre-market, explorative, early feasibility, pilot, controlled clinical investigation designed to collect initial clinical data on the medical device Previct Drugs.

DETAILED DESCRIPTION:
This first study will give valuable information on the feasibility of Previct Drugs function to measure pupils and eye movements and to evaluate if there are any changes in the pupillometric parameters before and after intake of a medicinal product. It will also provide information on the usability of the device. Drug intake will in this first investigation be simulated by a controlled single application of commonly therapeutically used medicinal products from the following classes of drugs: phenethylamines (D1), benzodiazepines (D2), cannabinoids (D3), and opioids (D4).

ELIGIBILITY:
Inclusion Criteria:

* Male or female healthy volunteers
* Age 18 to 70 years
* BMI between 18.5-30 kg/m2
* Weight between 50-100 kg
* Healthy as determined by the investigator or designee based on pre-study medical and surgical history and a health examination at enrollment
* Women of childbearing potential (defined as all women who are not surgically sterile or postmenopausal for at least 1 year prior to enrollment) must have a negative urine pregnancy test at enrollment and at visit 2 and must agree to use a medically acceptable contraception from enrollment until study completion
* No current drug usage defined as a negative urine drug test at enrollment and at visit 2
* Able to use Previct Drugs after initial training (defined as successfully performing a test after trying maximum three times per measurement)
* Been informed of the nature, the scope, and the relevance of the clinical investigation
* Voluntarily agreed on participation and has duly singed the Informed Consent Form

Exclusion Criteria:

* Participating in another clinical investigation which may affect the study outcome according to clinical judgement
* Pregnancy or Lactating
* Blind
* Deaf
* Abnormal ECG (QTc time >450 ms) at enrollment
* Current or recent history of alcohol misuse assessed by AUDIT where ≥6 points for women or ≥8 points for men indicates a potential misuse
* Current or history of psychiatric disorder or drug misuse assessed by M.I.N.I where the outcome will be based on clinical judgement
* Any disease or condition that may influence pupillary reflexes based on clinical judgement
* Undergone eye surgery that may influence pupillary reflexes based on clinical judgement
* Ongoing treatment with medications which may interfere with eye measurements based on clinical judgement
* Ongoing treatment with medications which may interfere with any of the medicinal products to be used
* History or presence of allergy or serious reaction to the medicinal products to be used
* History or presence of cardiovascular disease, e.g., arteriosclerosis, hypertension, or cor pulmonale
* History or presence of sleep-related breath disorder
* History or presence of gastrointestinal disease, e.g., paralytic ileus, acute abdomen, delayed gastric emptying, or chronic constipation
* History or presence of pulmonary disease, e.g., acute pulmonary insufficiency, severe respiratory depression with hypoxia, chronic obstructive lung disease, or bronchial asthma
* History or presence of autoimmune neuromuscular disease, e.g., myasthenia gravis
* Not able to read or understand the local language
* Any other condition that as judged by the investigator may make the follow-up or investigation inappropriate
* That according to the Declaration of Helsinki is deemed unsuitable for study enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markku Hämäläinen, PhD, Study Chair — Kontigo Care AB
Locations (1):
- Leiden University Medical Center (LUMC) Department of Anesthesiology, Leiden, Netherlands

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 48 subjects were included in the Full Analysis Set (FAS), 12 subjects per medicinal product type.
Groups:
- Healthy Volunteers With Single Application of Phenethylamines (D1): Evaluation of performance, safety, and usability of Previct Drugs when used in healthy volunteers allocated to one out of four medicinal products at Visit 2 to simulate drug use. Phenethylamines (D1) allocated to this specific group.
- Healthy Volunteers With Single Application of Benzodiazepines (D2): Evaluation of performance, safety, and usability of Previct Drugs when used in healthy volunteers allocated to one out of four medicinal products at Visit 2 to simulate drug use. Benzodiazepines (D2) allocated to this specific group.
- Healthy Volunteers With Single Application of Cannabinoids (D3): Evaluation of performance, safety, and usability of Previct Drugs when used in healthy volunteers allocated to one out of four medicinal products at Visit 2 to simulate drug use. Cannabinoids (D3) allocated to this specific group.
- Healthy Volunteers With Single Application of Opioids (D4): Evaluation of performance, safety, and usability of Previct Drugs when used in healthy volunteers allocated to one out of four medicinal products at Visit 2 to simulate drug use. Opioids (D4) allocated to this specific group.
Period: Overall Study
Arm/Group | Healthy Volunteers With Single Application of Phenethylamines (D1) | Healthy Volunteers With Single Application of Benzodiazepines (D2) | Healthy Volunteers With Single Application of Cannabinoids (D3) | Healthy Volunteers With Single Application of Opioids (D4)
Started | 12 | 12 | 12 | 12
Completed | 12 | 12 | 12 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS)
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteers With Single Application of Phenethylamines (D1) | Healthy Volunteers With Single Application of Benzodiazepines (D2) | Healthy Volunteers With Single Application of Cannabinoids (D3) | Healthy Volunteers With Single Application of Opioids (D4) | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.25 (12.90) | 27.92 (14.68) | 27.75 (17.35) | 28.00 (16.60) | 27.48 (15.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 7 | 8 | 34
  Male | 2 | 3 | 5 | 4 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Eye color [Count of Participants; unit: Participants]
  Eye color - blue | 7 | 2 | 7 | 8 | 24
  Eye color - grey | 2 | 0 | 1 | 0 | 3
  Eye color - green | 0 | 5 | 0 | 1 | 6
  Eye color - amber | 0 | 0 | 0 | 0 | 0
  Eye color - brown | 3 | 4 | 3 | 3 | 13
  Eye color - black | 0 | 0 | 0 | 0 | 0
  Eye color - other | 0 | 1 | 1 | 0 | 2
Audit questionnaire [Mean (Standard Deviation); unit: Score on a scale] — The audit questionnaire is assessing current or recent history of alcohol misuse and consists of 10 questions that each, depending on answer, gives the responder a score between 0 and 4 where higher scores corresponds to alcohol misuse. In total, the person completing the audit questionnaire can get a score between 0 and 40.
  Score on a scale | 4.42 (1.08) | 3.83 (2.12) | 4.5 (2.11) | 5.08 (1.62) | 4.46 (1.79)

OUTCOME MEASURES:

1. Primary Outcome: Use of Self-administered Pupillometry Using a Mobile Phone Application Can be Used to Collect Pupillograms Before and Under the Influence of Phenethylamines, Benzodiazepines, Cannabinoids, and Opioids (D1-D4).
Description: For each medicinal product (D1-D4), the fraction of collected pupillometry data from the mobile phone application at baseline and under the influence of D1-D4, which can be transformed into pre-defined key features using native pupillogram. A key feature represents an eye characteristic (such as pupil size, iris position, and the similar). A successful transformation is characterised by underlying quality control algorithms approving the extracted magnitude, where poor quality pupillograms are rejected from analysis. Each attempt to transform a pupillogram into key features is denoted an "Attempt", and the successful transformation is denoted a "Successful attempt".
Time Frame: Day 7 +/- 2 days (Visit 2)
Population: FAS population. Participating subjects were allowed to have several attempts per test if needed. Consequently the number of analyzed attempts differ between groups and also between the different test types (NC, NY, TR, PLR, RED).
Measure: Count of Units; unit: Number of attempts
Units Other Than Participants: Number of attempts
Arm/Group | Single Application of Phenethylamines (D1) | Single Application of Benzodiazepines (D2) | Single Application of Cannabinoids (D3) | Single Application of Opioids (D4)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Number analyzed (Number of attempts) | 320 | 329 | 339 | 336
Number of attempts
  Successful attempts - Non-convergence (NC): number analyzed (Number of attempts) | 309 | 295 | 339 | 332
  Successful attempts - Non-convergence (NC) | 295 | 286 | 317 | 300
  Successful attempts - Horizontal nystagmus (NY): number analyzed (Number of attempts) | 312 | 307 | 333 | 318
  Successful attempts - Horizontal nystagmus (NY) | 279 | 242 | 300 | 282
  Successful attempts - Tremor (TR): number analyzed (Number of attempts) | 312 | 307 | 333 | 318
  Successful attempts - Tremor (TR) | 295 | 282 | 319 | 295
  Successful attempts - Pupillary light reflex (PLR): number analyzed (Number of attempts) | 320 | 329 | 321 | 336
  Successful attempts - Pupillary light reflex (PLR) | 290 | 297 | 302 | 307
  Successful attempts - Redness (RED): number analyzed (Number of attempts) | 320 | 329 | 321 | 336
  Successful attempts - Redness (RED) | 314 | 317 | 312 | 325

2. Secondary Outcome: Use of Self-administered Pupillometry Using a Mobile Phone Application, After Refining the Method for Establishing Pupillograms, Can be Used to Collect Pupillograms Before and Under the Influence of Each Medicinal Product (D1-D4).
Description: For each medicinal product (D1-D4), the fraction of collected pupillometry data from the mobile phone application at baseline and under the influence of D1-D4, which can be transformed into pre-defined key features using refined pupillogram. A key feature represents an eye characteristic (such as pupil size, iris position, and the similar). A successful transformation is characterised by underlying quality control algorithms approving the extracted magnitude, where poor quality pupillograms are rejected from analysis. Each attempt to transform a pupillogram into key features is denoted an "Attempt", and the successful transformation is denoted a "Successful attempt.
Time Frame: Day 7 +/- 2 days (Visit 2)
Population: as for outcome 1
Measure: Count of Units; unit: Successful attempts
Units Other Than Participants: Successful attempts
Arm/Group | Single Application of Phenethylamines (D1) | Single Application of Benzodiazepines (D2) | Single Application of Cannabinoids (D3) | Single Application of Opioids (D4)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Number analyzed (Successful attempts) | 320 | 329 | 339 | 336
Successful attempts
  Successful attempts - Non-convergence (NC): number analyzed (Successful attempts) | 309 | 295 | 339 | 332
  Successful attempts - Non-convergence (NC) | 296 | 282 | 318 | 297
  Successful attempts - Horizontal nystagmus (NY): number analyzed (Successful attempts) | 312 | 307 | 333 | 318
  Successful attempts - Horizontal nystagmus (NY) | 281 | 241 | 305 | 281
  Successful attempts - Tremor (TR): number analyzed (Successful attempts) | 312 | 307 | 333 | 318
  Successful attempts - Tremor (TR) | 295 | 282 | 319 | 295
  Successful attempts - Pupillary light reflex (PLR): number analyzed (Successful attempts) | 320 | 329 | 321 | 336
  Successful attempts - Pupillary light reflex (PLR) | 294 | 303 | 309 | 317
  Successful attempts - Redness (RED): number analyzed (Successful attempts) | 320 | 329 | 321 | 336
  Successful attempts - Redness (RED) | 314 | 317 | 312 | 325

3. Secondary Outcome: Number of Key Features With Change From Baseline to Peak Concentration in Plasma, Using Refined Pupillograms.
Description: For each medicinal product (D1-D4), number of changed key features from baseline to the LC-MS/MS (Liquid Chromatography Tandem Mass-Spectroscopy) verified peak concentration in plasma after administration of medicinal product at visit 2 using refined pupillograms. Each of the 24 key features represents an eye characteristic (such as pupil size, iris position, and the similar). A key feature is considered "changed" if the difference between averages at baseline and peak concentration is significant (p<0.05). Key features were available from two conditions, one condition where pupillograms and corresponding key features were collected in dim ambient light (50 Lux) and one condition where pupillograms and corresponding key features were collected in bright ambient light (500 Lux). The Outcome Measure is reported for both ambient light conditions.
Time Frame: Day 7 +/- 2 days (Visit 2)
Population: FAS population.
Measure: Count of Units; unit: Number of key features
Units Other Than Participants: Number of key features
Groups:
- Single Application of Phenethylamines: Evaluation of Previct Drugs' function to measure pupils and eye movements and to evaluate if there are any changes in the pupillometric parameters before and after intake of phenethylamines.
- Single Application of Benzodiazepines: Evaluation of Previct Drugs' function to measure pupils and eye movements and to evaluate if there are any changes in the pupillometric parameters before and after intake of benzodiazepines.
- Single Application of Cannabinoids: Evaluation of Previct Drugs' function to measure pupils and eye movements and to evaluate if there are any changes in the pupillometric parameters before and after intake of cannabinoids.
- Single Application of Opioids: Evaluation of Previct Drugs' function to measure pupils and eye movements and to evaluate if there are any changes in the pupillometric parameters before and after intake of opioids.
Arm/Group | Single Application of Phenethylamines | Single Application of Benzodiazepines | Single Application of Cannabinoids | Single Application of Opioids
Number analyzed (Participants) | 12 | 12 | 12 | 12
Number analyzed (Number of key features) | 24 | 24 | 24 | 24
Number of key features
  50 Lux | 5 | 1 | 4 | 7
  500 Lux | 5 | 3 | 2 | 7

4. Secondary Outcome: Number of Key Features for Which Correlation Between Pupillometric Variables and Concentration in Plasma Over Time is Significant for Each Medicinal Product D1-D4 and Ambient Light Condition.
Description: For each medicinal product (D1-D4), number of significant correlations between key features and plasma concentration over time using refined pupillograms. A key feature represents an eye characteristic (such as pupil size, iris position, and the similar). A key feature is considered "correlated" if the slope in a linear regression is significantly different from zero (p<0.05). The term correlated over time refers to data collected during 5 hours at Visit 2 after administration of D1-D4. Key features were available from two conditions, one condition where pupillograms and corresponding key features were collected in dim ambient light (50 Lux) and one condition where pupillograms and corresponding key features were collected in bright ambient light (500 Lux). The Outcome Measure is reported for both ambient light conditions.
Time Frame: Day 7 +/- 2 days (Visit 2)
Population: FAS population.
Measure: Count of Units; unit: Number of key features
Units Other Than Participants: Number of key features
Arm/Group | Single Application of Phenethylamines | Single Application of Benzodiazepines | Single Application of Cannabinoids | Single Application of Opioids
Number analyzed (Participants) | 12 | 12 | 12 | 12
Number analyzed (Number of key features) | 24 | 24 | 24 | 24
Number of key features
  50 LUX | 5 | 6 | 7 | 10
  500 LUX | 7 | 4 | 2 | 9
Statistical Analysis 1: Comparison: Single Application of Phenethylamines; The correlation between pupillometric variables and concentration in plasma over time for designated medicinal product and ambient light condition was evaluated by collecting all pairs of (key feature value) and (plasma concentration). For each key feature, medicinal product, and ambient light condition, a linear regression was conducted producing an estimate of k and m in the following equation (key feature value) = k * (plasma concentration) + m; Test type: Other — The hypothesis was that k = 0. If the hypothesis could be rejected (p<0.05), then the pupillometric variable was considered correlated with plasma concentration for the particular key feature, medicinal product and ambient light condition. Here the p-value for Dbase at 50 lux is reported; p < 0.0001, Regression, Linear; Slope = 7.11
Statistical Analysis 2: Comparison: Single Application of Phenethylamines; [analysis description as in outcome 4, analysis 1]; Test type: Other — The hypothesis was that k = 0. If the hypothesis could be rejected (p<0.05), then the pupillometric variable was considered correlated with plasma concentration for the particular key feature, medicinal product and ambient light condition. Here the p-value for Dcon at 50 lux is reported; p < 0.0001, Regression, Linear; Slope = 5.98
Statistical Analysis 3: Comparison: Single Application of Phenethylamines; [analysis description as in outcome 4, analysis 1]; Test type: Other — The hypothesis was that k = 0. If the hypothesis could be rejected (p<0.05), then the pupillometric variable was considered correlated with plasma concentration for the particular key feature, medicinal product and ambient light condition. Here the p-value for Ctime at 50 lux is reported; p = 0.0006, Regression, Linear; Slope = 7.17
Statistical Analysis 4: Comparison: Single Application of Phenethylamines; [analysis description as in outcome 4, analysis 1]; Test type: Other — The hypothesis was that k = 0. If the hypothesis could be rejected (p<0.05), then the pupillometric variable was considered correlated with plasma concentration for the particular key feature, medicinal product and ambient light condition. Here the p-value for Dend at 50 lux is reported; p < 0.0001, Regression, Linear; Slope = 4.75
Statistical Analysis 5: Comparison: Single Application of Phenethylamines; [analysis description as in outcome 4, analysis 1]; Test type: Other — The hypothesis was that k = 0. If the hypothesis could be rejected (p<0.05), then the pupillometric variable was considered correlated with plasma concentration for the particular key feature, medicinal product and ambient light condition. Here the p-value for MCA at 50 lux is reported; p = 0.0002, Regression, Linear; Slope = 5.95
Statistical Analysis 6: Comparison: Single Application of Phenethylamines; [analysis description as in outcome 4, analysis 1]; Test type: Other — The hypothesis was that k = 0. If the hypothesis could be rejected (p<0.05), then the pupillometric variable was considered correlated with plasma concentration for the particular key feature, medicinal product and ambient light condition. Here the p-value for D2m at 500 lux is reported; p = 0.0285, Regression, Linear; Slope = 6.92
Statistical Analysis 7: Comparison: Single Application of Phenethylamines; [analysis description as in outcome 4, analysis 1]; Test type: Other — The hypothesis was that k = 0. If the hypothesis could be rejected (p<0.05), then the pupillometric variable was considered correlated with plasma concentration for the particular key feature, medicinal product and ambient light condition. Here the p-value for Dbase at 500 lux is reported; p < 0.0001, Regression, Linear; Slope = 6.99
Statistical Analysis 8: Comparison: Single Application of Phenethylamines; [analysis description as in outcome 4, analysis 1]; Test type: Other — The hypothesis was that k = 0. If the hypothesis could be rejected (p<0.05), then the pupillometric variable was considered correlated with plasma concentration for the particular key feature, medicinal product and ambient light condition. Here the p-value for Dcon at 500 lux is reported; p < 0.0001, Regression, Linear; Slope = 6.8
Statistical Analysis 9: Comparison: Single Application of Phenethylamines; [analysis description as in outcome 4, analysis 1]; Test type: Other — The hypothesis was that k = 0. If the hypothesis could be rejected (p<0.05), then the pupillometric variable was considered correlated with plasma concentration for the particular key feature, medicinal product and ambient light condition. Here the p-value for Dend at 500 lux is reported; p = 0.0001, Regression, Linear; Slope = 5.94
Statistical Analysis 10: Comparison: Single Application of Phenethylamines; [analysis description as in outcome 4, analysis 1]; Test type: Other — The hypothesis was that k = 0. If the hypothesis could be rejected (p<0.05), then the pupillometric variable was considered correlated with plasma concentration for the particular key feature, medicinal product and ambient light condition. Here the p-value for MCA at 500 lux is reported; p = 0.012, Regression, Linear; Slope = 5.85
Statistical Analysis 11: Comparison: Single Application of Phenethylamines; [analysis description as in outcome 4, analysis 1]; Test type: Other — The hypothesis was that k = 0. If the hypothesis could be rejected (p<0.05), then the pupillometric variable was considered correlated with plasma concentration for the particular key feature, medicinal product and ambient light condition. Here the p-value for NYmass at 500 lux is reported; p = 0.0174, Regression, Linear; Slope = -9.62
Statistical Analysis 12: Comparison: Single Application of Phenethylamines; [analysis description as in outcome 4, analysis 1]; Test type: Other — The hypothesis was that k = 0. If the hypothesis could be rejected (p<0.05), then the pupillometric variable was considered correlated with plasma concentration for the particular key feature, medicinal product and ambient light condition. Here the p-value for D1m at 500 lux is reported; p = 0.013, Regression, Linear; Slope = -9.15
Statistical Analysis 13: Comparison: Single Application of Benzodiazepines; [analysis description as in outcome 4, analysis 1]; Test type: Other — The hypothesis was that k = 0. If the hypothesis could be rejected (p<0.05), then the pupillometric variable was considered correlated with plasma concentration for the particular key feature, medicinal product and ambient light condition. Here the p-value for NCdiff at 50 lux is reported; p < 0.0001, Regression, Linear; Slope = -4.06
Statistical Analysis 14: Comparison: Single Application of Benzodiazepines; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 1]; p = 0.0068, Regression, Linear; Slope = 0.99
Statistical Analysis 15: Comparison: Single Application of Benzodiazepines; [analysis description as in outcome 4, analysis 1]; Test type: Other — The hypothesis was that k = 0. If the hypothesis could be rejected (p<0.05), then the pupillometric variable was considered correlated with plasma concentration for the particular key feature, medicinal product and ambient light condition. Here the p-value for MCV at 50 lux is reported; p = 0.0485, Regression, Linear; Slope = 1.12
Statistical Analysis 16: Comparison: Single Application of Benzodiazepines; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 3]; p = 0.0031, Regression, Linear; Slope = 2.08
Statistical Analysis 17: Comparison: Single Application of Benzodiazepines; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 5]; p = 0.0036, Regression, Linear; Slope = 1.18
Statistical Analysis 18: Comparison: Single Application of Benzodiazepines; [analysis description as in outcome 4, analysis 1]; Test type: Other — The hypothesis was that k = 0. If the hypothesis could be rejected (p<0.05), then the pupillometric variable was considered correlated with plasma concentration for the particular key feature, medicinal product and ambient light condition. Here the p-value for RMCA at 50 lux is reported; p = 0.0089, Regression, Linear; Slope = 1.05
Statistical Analysis 19: Comparison: Single Application of Benzodiazepines; [analysis description as in outcome 4, analysis 1]; Test type: Other — The hypothesis was that k = 0. If the hypothesis could be rejected (p<0.05), then the pupillometric variable was considered correlated with plasma concentration for the particular key feature, medicinal product and ambient light condition. Here the p-value for NCdiff at 500 lux is reported; p < 0.0001, Regression, Linear; Slope = -4.04
Statistical Analysis 20: Comparison: Single Application of Benzodiazepines; [analysis description as in outcome 4, analysis 1]; Test type: Other — The hypothesis was that k = 0. If the hypothesis could be rejected (p<0.05), then the pupillometric variable was considered correlated with plasma concentration for the particular key feature, medicinal product and ambient light condition. Here the p-value for MM30 at 500 lux is reported; p = 0.0239, Regression, Linear; Slope = 1.62
Statistical Analysis 21: Comparison: Single Application of Benzodiazepines; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 8]; p = 0.0435, Regression, Linear; Slope = 0.93
Statistical Analysis 22: Comparison: Single Application of Benzodiazepines; [analysis description as in outcome 4, analysis 1]; Test type: Other — The hypothesis was that k = 0. If the hypothesis could be rejected (p<0.05), then the pupillometric variable was considered correlated with plasma concentration for the particular key feature, medicinal product and ambient light condition. Here the p-value for Ctime at 500 lux is reported; p = 0.0126, Regression, Linear; Slope = 1.26
Statistical Analysis 23: Comparison: Single Application of Cannabinoids; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 13]; p = 0.0294, Regression, Linear; Slope = -0.73
Statistical Analysis 24: Comparison: Single Application of Cannabinoids; [analysis description as in outcome 4, analysis 1]; Test type: Other — The hypothesis was that k = 0. If the hypothesis could be rejected (p<0.05), then the pupillometric variable was considered correlated with plasma concentration for the particular key feature, medicinal product and ambient light condition. Here the p-value for D1m at 50 lux is reported; p = 0.0204, Regression, Linear; Slope = 0.96
Statistical Analysis 25: Comparison: Single Application of Cannabinoids; [analysis description as in outcome 4, analysis 1]; Test type: Other — The hypothesis was that k = 0. If the hypothesis could be rejected (p<0.05), then the pupillometric variable was considered correlated with plasma concentration for the particular key feature, medicinal product and ambient light condition. Here the p-value for D2m at 50 lux is reported; p = 0.0004, Regression, Linear; Slope = 1.41
Statistical Analysis 26: Comparison: Single Application of Cannabinoids; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 15]; p = 0.0013, Regression, Linear; Slope = -0.95
Statistical Analysis 27: Comparison: Single Application of Cannabinoids; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 5]; p = 0.0003, Regression, Linear; Slope = -0.77
Statistical Analysis 28: Comparison: Single Application of Cannabinoids; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 18]; p < 0.0001, Regression, Linear; Slope = -0.94
Statistical Analysis 29: Comparison: Single Application of Cannabinoids; [analysis description as in outcome 4, analysis 1]; Test type: Other — The hypothesis was that k = 0. If the hypothesis could be rejected (p<0.05), then the pupillometric variable was considered correlated with plasma concentration for the particular key feature, medicinal product and ambient light condition. Here the p-value for Redness at 50 lux is reported; p < 0.0001, Regression, Linear; Slope = 0.81
Statistical Analysis 30: Comparison: Single Application of Cannabinoids; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 19]; p = 0.0096, Regression, Linear; Slope = -0.87
Statistical Analysis 31: Comparison: Single Application of Cannabinoids; [analysis description as in outcome 4, analysis 1]; Test type: Other — The hypothesis was that k = 0. If the hypothesis could be rejected (p<0.05), then the pupillometric variable was considered correlated with plasma concentration for the particular key feature, medicinal product and ambient light condition. Here the p-value for Redness at 500 lux is reported; p = 0.0003, Regression, Linear; Slope = 0.36
Statistical Analysis 32: Comparison: Single Application of Opioids; [analysis description as in outcome 4, analysis 1]; Test type: Other — The hypothesis was that k = 0. If the hypothesis could be rejected (p<0.05), then the pupillometric variable was considered correlated with plasma concentration for the particular key feature, medicinal product and ambient light condition. Here the p-value for MM10 at 50 lux is reported; p = 0.0063, Regression, Linear; Slope = 2.13
Statistical Analysis 33: Comparison: Single Application of Opioids; [analysis description as in outcome 4, analysis 1]; Test type: Other — The hypothesis was that k = 0. If the hypothesis could be rejected (p<0.05), then the pupillometric variable was considered correlated with plasma concentration for the particular key feature, medicinal product and ambient light condition. Here the p-value for MM30 at 50 lux is reported; p = 0.0018, Regression, Linear; Slope = 2.30
Statistical Analysis 34: Comparison: Single Application of Opioids; [analysis description as in outcome 4, analysis 1]; Test type: Other — The hypothesis was that k = 0. If the hypothesis could be rejected (p<0.05), then the pupillometric variable was considered correlated with plasma concentration for the particular key feature, medicinal product and ambient light condition. Here the p-value for Pa at 50 lux is reported; p = 0.0134, Regression, Linear; Slope = 3.22
Statistical Analysis 35: Comparison: Single Application of Opioids; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 1]; p < 0.0001, Regression, Linear; Slope = -1.48
Statistical Analysis 36: Comparison: Single Application of Opioids; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 15]; p < 0.0001, Regression, Linear; Slope = -2.48
Statistical Analysis 37: Comparison: Single Application of Opioids; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 2]; p < 0.0001, Regression, Linear; Slope = -1.264
Statistical Analysis 38: Comparison: Single Application of Opioids; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 4]; p < 0.0001, Regression, Linear; Slope = -1.47
Statistical Analysis 39: Comparison: Single Application of Opioids; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 5]; p < 0.0001, Regression, Linear; Slope = -1.64
Statistical Analysis 40: Comparison: Single Application of Opioids; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 18]; p < 0.0001, Regression, Linear; Slope = -1.63
Statistical Analysis 41: Comparison: Single Application of Opioids; [analysis description as in outcome 4, analysis 1]; Test type: Other — The hypothesis was that k = 0. If the hypothesis could be rejected (p<0.05), then the pupillometric variable was considered correlated with plasma concentration for the particular key feature, medicinal product and ambient light condition. Here the p-value for PESC at 50 lux is reported; p = 0.0313, Regression, Linear; Slope = 1.43
Statistical Analysis 42: Comparison: Single Application of Opioids; [analysis description as in outcome 4, analysis 1]; Test type: Other — The hypothesis was that k = 0. If the hypothesis could be rejected (p<0.05), then the pupillometric variable was considered correlated with plasma concentration for the particular key feature, medicinal product and ambient light condition. Here the p-value for MM5 at 500 lux is reported; p = 0.0481, Regression, Linear; Slope = 1.92
Statistical Analysis 43: Comparison: Single Application of Opioids; [analysis description as in outcome 4, analysis 1]; Test type: Other — The hypothesis was that k = 0. If the hypothesis could be rejected (p<0.05), then the pupillometric variable was considered correlated with plasma concentration for the particular key feature, medicinal product and ambient light condition. Here the p-value for MM10 at 500 lux is reported; p = 0.0171, Regression, Linear; Slope = 2.57
Statistical Analysis 44: Comparison: Single Application of Opioids; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 20]; p = 0.0007, Regression, Linear; Slope = 3.84
Statistical Analysis 45: Comparison: Single Application of Opioids; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 7]; p < 0.0001, Regression, Linear; Slope = -2.15
Statistical Analysis 46: Comparison: Single Application of Opioids; [analysis description as in outcome 4, analysis 1]; Test type: Other — The hypothesis was that k = 0. If the hypothesis could be rejected (p<0.05), then the pupillometric variable was considered correlated with plasma concentration for the particular key feature, medicinal product and ambient light condition. Here the p-value for MCV at 500 lux is reported; p < 0.0001, Regression, Linear; Slope = -2.20
Statistical Analysis 47: Comparison: Single Application of Opioids; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 8]; p < 0.0001, Regression, Linear; Slope = -2.44
Statistical Analysis 48: Comparison: Single Application of Opioids; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 9]; p < 0.0001, Regression, Linear; Slope = -3.01
Statistical Analysis 49: Comparison: Single Application of Opioids; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 10]; p < 0.0001, Regression, Linear; Slope = -1.82
Statistical Analysis 50: Comparison: Single Application of Opioids; [analysis description as in outcome 4, analysis 1]; Test type: Other — The hypothesis was that k = 0. If the hypothesis could be rejected (p<0.05), then the pupillometric variable was considered correlated with plasma concentration for the particular key feature, medicinal product and ambient light condition. Here the p-value for RMCA at 500 lux is reported; p < 0.0001, Regression, Linear; Slope = -1.83

5. Secondary Outcome: Number of Key Features With Change From Baseline to 5 Hours After Administration of Medicinal Product, Using Refined Pupillograms.
Description: For each medicinal product (D1-D4), number of changed key features from baseline to 5 hours after administration of medicinal product at visit 2 using refined pupillograms. A key feature represents an eye characteristic (such as pupil size, iris position, and the similar). A key feature is considered "changed" if the difference between averages at baseline and at 5 hours is significant (p<0.05). Key features were available from two conditions, one condition where pupillograms and corresponding key features were collected in dim ambient light (50 Lux) and one condition where pupillograms and corresponding key features were collected in bright ambient light (500 Lux). The Outcome Measure is reported for both ambient light conditions.
Time Frame: Day 7 +/- 2 days (Visit 2)
Population: FAS population.
Measure: Count of Units; unit: Number of Key features
Units Other Than Participants: Number of Key features
Arm/Group | Single Application of Phenethylamines | Single Application of Benzodiazepines | Single Application of Cannabinoids | Single Application of Opioids
Number analyzed (Participants) | 12 | 12 | 12 | 12
Number analyzed (Number of Key features) | 24 | 24 | 24 | 24
Number of Key features
  50 LUX | 6 | 1 | 2 | 8
  500 LUX | 5 | 5 | 0 | 6

6. Secondary Outcome: Number of Correct Classifications of Subjects, Evaluated Using a Combination of Different Pupillometric Variables for Indicating Use of Each Medicinal Product D1-D4 and Ambient Light Condition.
Description: For each medicinal product (D1-D4), evaluate known combinations of key features that changes from baseline to the LC-MS/MS verified peak concentration in plasma after administration of medicinal product at visit 2 using refined pupillograms. A key feature represents an eye characteristic (such as pupil size, iris position, and the similar). A combination of key features collected at peak plasma concentration was used to build a logistic regression classifier, and the resulting counts of true positives, true negatives, false positives, and false negatives are presented. Key features were available from two conditions, one condition where pupillograms and corresponding key features were collected in dim ambient light (50 Lux) and one condition where pupillograms and corresponding key features were collected in bright ambient light (500 Lux). The Outcome Measure is reported for both ambient light conditions. Key feature values were missing in a few instances, as shown in the table.
Time Frame: Day 7 +/- 2 days (Visit 2)
Population: FAS population. Obtained measurement data included for all subjects where available. Data for 500 Lux Kay feature Dbase missing for one subject in group D4 (opioid group). Consequently, data from 11 subjects presented for this variable.
Measure: Number; unit: Number of participants
Groups:
- Single Application of Phenethylamines - 50 Lux Key Feature Dbase; Single Application of Phenethylamines - 500 Lux Key Feature Dbase: Evaluation of Previct Drugs' function to measure pupils and eye movements and to evaluate if there are any changes in the pupillometric parameters before and after intake of phenethylamines.
- Single Application of Benzodiazepines - 50 Lux Key Feature NCdiff; Single Application of Benzodiazepines - 500 Lux Key Feature NCdiff; Single Application of Benzodiazepines - 500 Lux Key Feature NCdiff-NYave: Evaluation of Previct Drugs' function to measure pupils and eye movements and to evaluate if there are any changes in the pupillometric parameters before and after intake of benzodiazepines.
- Single Application of Cannabinoids - 50 Lux Key Feature MCA; Single Application of Cannabinoids - 50 Lux Key Feature MCA + Redness; Single Application of Cannabinoids - 500 Lux Key Feature Redness; Single Application of Cannabinoids - 500 Lux Key Feature Redness+NYNumber: Evaluation of Previct Drugs' function to measure pupils and eye movements and to evaluate if there are any changes in the pupillometric parameters before and after intake of cannabinoids.
- Single Application of Opioids - 50 Lux Key Feature Dbase; Single Application of Opioids - 500 Lux Key Feature Dbase: Evaluation of Previct Drugs' function to measure pupils and eye movements and to evaluate if there are any changes in the pupillometric parameters before and after intake of opioids.
Arm/Group | Single Application of Phenethylamines - 50 Lux Key Feature Dbase | Single Application of Phenethylamines - 500 Lux Key Feature Dbase | Single Application of Benzodiazepines - 50 Lux Key Feature NCdiff | Single Application of Benzodiazepines - 500 Lux Key Feature NCdiff | Single Application of Benzodiazepines - 500 Lux Key Feature NCdiff-NYave | Single Application of Cannabinoids - 50 Lux Key Feature MCA | Single Application of Cannabinoids - 50 Lux Key Feature MCA + Redness | Single Application of Cannabinoids - 500 Lux Key Feature Redness | Single Application of Cannabinoids - 500 Lux Key Feature Redness+NYNumber | Single Application of Opioids - 50 Lux Key Feature Dbase | Single Application of Opioids - 500 Lux Key Feature Dbase
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Number of participants
  At baseline number of true negative: number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 11
  At baseline number of true negative | 12 | 12 | 12 | 10 | 11 | 12 | 12 | 12 | 11 | 12 | 11
  At baseline number of false positive: number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 11
  At baseline number of false positive | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  At baseline, missing key feature data | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  At peak concentration number of true positive: number analyzed (Participants) | 12 | 12 | 12 | 12 | 11 | 11 | 11 | 11 | 10 | 12 | 11
  At peak concentration number of true positive | 12 | 12 | 12 | 11 | 10 | 10 | 11 | 8 | 9 | 12 | 11
  At peak concentration number of false negative: number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 11
  At peak concentration number of false negative | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 3 | 1 | 0 | 0
  At peak concentration, missing key feature data | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 1
Statistical Analysis 1: Comparison: Single Application of Phenethylamines - 50 Lux Key Feature Dbase vs Single Application of Phenethylamines - 500 Lux Key Feature Dbase vs Single Application of Benzodiazepines - 50 Lux Key Feature NCdiff vs Single Application of Opioids - 50 Lux Key Feature Dbase; The null hypothesis is that the logistic regression classifier is unable to correctly classify subjects into sober or under the influence of D1-D4. The smallest odds ratio from the group false positives and false negative is reported; Test type: Other; p < 0.05, Regression, Logistic; probability = 0.000244
Statistical Analysis 2: Comparison: Single Application of Benzodiazepines - 500 Lux Key Feature NCdiff-NYave vs Single Application of Cannabinoids - 50 Lux Key Feature MCA; The null hypothesis is that the logistic regression classifier is unable to correctly classify subjects into sober or under the influence of D1-D4. The greatest p value from the group false positives and false negative is reported; Test type: Other; p < 0.05, Regression, Logistic; probability = 0.00586
Statistical Analysis 3: Comparison: Single Application of Benzodiazepines - 500 Lux Key Feature NCdiff; [analysis description as in outcome 6, analysis 2]; Test type: Other; p < 0.05, Regression, Logistic; probability = 0.0193
Statistical Analysis 4: Comparison: Single Application of Cannabinoids - 50 Lux Key Feature MCA + Redness vs Single Application of Opioids - 500 Lux Key Feature Dbase; [analysis description as in outcome 6, analysis 2]; Test type: Other; p < 0.05, Regression, Logistic; probability = 0.000488
Statistical Analysis 5: Comparison: Single Application of Cannabinoids - 500 Lux Key Feature Redness; [analysis description as in outcome 6, analysis 2]; Test type: Other; p < 0.05, Regression, Logistic; probability = 0.1133
Statistical Analysis 6: Comparison: Single Application of Cannabinoids - 500 Lux Key Feature Redness+NYNumber; Test type: Other; p < 0.05, Regression, Logistic; probability = 0.0107

7. Secondary Outcome: Usability Questionnaire - Question 1
Description: User-friendliness of Previct Drugs evaluated by the subject at visit 2. Question 1. How would you grade the instructions for use?
  Response options:
  * Not understandable
  * Could only understand some parts
  * Could understand most parts
  * Could understand almost every part
  * Fully understandable
Time Frame: Day 7 +/- 2 days (Visit 2)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers With Single Application of Phenethylamines (D1) | Healthy Volunteers With Single Application of Benzodiazepines (D2) | Healthy Volunteers With Single Application of Cannabinoids (D3) | Healthy Volunteers With Single Application of Opioids (D4)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  Not understandable | 0 | 0 | 0 | 0
  Could only understand some parts | 0 | 0 | 0 | 0
  Could understand most parts | 0 | 1 | 0 | 0
  Could understand almost every part | 1 | 5 | 5 | 3
  Fully understandable | 11 | 6 | 7 | 9

8. Secondary Outcome: Usability Questionnaire - Question 2
Description: User-friendliness of Previct Drugs evaluated by the subject at visit 2. Question 2. Was Previct Drugs easy to use correctly based on the information in the Instructions For Use (IFU)?
  Response options:
  * Yes
  * No
Time Frame: Day 7 +/- 2 days (Visit 2)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers With Single Application of Phenethylamines (D1) | Healthy Volunteers With Single Application of Benzodiazepines (D2) | Healthy Volunteers With Single Application of Cannabinoids (D3) | Healthy Volunteers With Single Application of Opioids (D4)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  Yes | 11 | 12 | 12 | 12
  No | 1 | 0 | 0 | 0

9. Secondary Outcome: Usability Questionnaire - Question 4
Description: User-friendliness of Previct Drugs evaluated by the subject at visit 2. Question 4. How did you experience the verbal instructions during a test with Previct Drugs?
  Response options:
  * Very easy to understand
  * Easy to understand
  * Nor easy or difficult to understand
  * Difficult to understand
  * Very difficult to understand
Time Frame: Day 7 +/- 2 days (Visit 2)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers With Single Application of Phenethylamines (D1) | Healthy Volunteers With Single Application of Benzodiazepines (D2) | Healthy Volunteers With Single Application of Cannabinoids (D3) | Healthy Volunteers With Single Application of Opioids (D4)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  Very easy to understand | 11 | 8 | 5 | 6
  Easy to understand | 1 | 4 | 7 | 6
  Nor easy or difficult to understand | 0 | 0 | 0 | 0
  Difficult to understand | 0 | 0 | 0 | 0
  Very difficult to understand | 0 | 0 | 0 | 0

10. Secondary Outcome: Usability Questionnaire - Question 5
Description: User-friendliness of Previct Drugs evaluated by the subject at visit 2. Question 5. Before starting a test, the App prompted you with a few written instructions. Did you read the instructions?
  Response options:
  * Yes
  * No
Time Frame: Day 7 +/- 2 days (Visit 2)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers With Single Application of Phenethylamines (D1) | Healthy Volunteers With Single Application of Benzodiazepines (D2) | Healthy Volunteers With Single Application of Cannabinoids (D3) | Healthy Volunteers With Single Application of Opioids (D4)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  Yes | 12 | 10 | 9 | 11
  No | 0 | 2 | 3 | 1

11. Secondary Outcome: Usability Questionnaire - Question 7
Description: User-friendliness of Previct Drugs evaluated by the subject at visit 2. Question 7. How did you experience performing a test with Previct Drugs (from opening of the App until the test was completed)?
  Response options:
  * Very easy to perform
  * Easy to perform
  * Nor easy or difficult to perform
  * Difficult to perform
  * Very difficult to perform
Time Frame: Day 7 +/- 2 days (Visit 2)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers With Single Application of Phenethylamines (D1) | Healthy Volunteers With Single Application of Benzodiazepines (D2) | Healthy Volunteers With Single Application of Cannabinoids (D3) | Healthy Volunteers With Single Application of Opioids (D4)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  Very easy to perform | 5 | 5 | 5 | 4
  Easy to perform | 7 | 5 | 5 | 8
  Nor easy or difficult to perform | 0 | 2 | 2 | 0
  Difficult to perform | 0 | 0 | 0 | 0
  Very difficult to perform | 0 | 0 | 0 | 0

12. Secondary Outcome: Usability Questionnaire - Question 8
Description: User-friendliness of Previct Drugs evaluated by the subject at visit 2. Question 8. During a test with Previct Drugs, did you at any time have to tilt the mobile against something to be able to perform a measurement?
  Response options:
  * Yes
  * No
Time Frame: Day 7 +/- 2 days (Visit 2)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers With Single Application of Phenethylamines (D1) | Healthy Volunteers With Single Application of Benzodiazepines (D2) | Healthy Volunteers With Single Application of Cannabinoids (D3) | Healthy Volunteers With Single Application of Opioids (D4)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  Yes | 4 | 3 | 4 | 4
  No | 8 | 9 | 8 | 8

13. Secondary Outcome: Usability Questionnaire - Question 9
Description: User-friendliness of Previct Drugs evaluated by the subject at visit 2.
  Question 9. If Yes (to question 8), how often did you have to tilt the mobile against something:
  Response options:
  * One occasion
  * Several occasions
  * Most occasions
  * All occasions
Time Frame: Day 7 +/- 2 days (Visit 2)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers With Single Application of Phenethylamines (D1) | Healthy Volunteers With Single Application of Benzodiazepines (D2) | Healthy Volunteers With Single Application of Cannabinoids (D3) | Healthy Volunteers With Single Application of Opioids (D4)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  One occasion | 1 | 2 | 2 | 1
  Several occasions | 3 | 1 | 2 | 3
  Most occasions | 0 | 0 | 0 | 0
  All occasions | 0 | 0 | 0 | 0
  Missing | 8 | 9 | 8 | 8

14. Secondary Outcome: Usability Questionnaire - Question 10
Description: User-friendliness of Previct Drugs evaluated by the subject at visit 2. Question 10. According to you, how many minutes did a test with Previct Drugs take in general? From start to end.
  Response options:
  * < 5 minutes
  * 5-7 minutes
  * > 7 minutes
Time Frame: Day 7 +/- 2 days (Visit 2)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers With Single Application of Phenethylamines (D1) | Healthy Volunteers With Single Application of Benzodiazepines (D2) | Healthy Volunteers With Single Application of Cannabinoids (D3) | Healthy Volunteers With Single Application of Opioids (D4)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  < 5 minutes | 5 | 2 | 3 | 2
  5-7 minutes | 5 | 6 | 4 | 7
  > 7 minutes | 2 | 4 | 5 | 3

15. Secondary Outcome: Usability Questionnaire - Question 11
Description: User-friendliness of Previct Drugs evaluated by the subject at visit 2. Question 11. Did you receive a notification when it was time for a test with Previct Drugs?
  Response options:
  * Yes
  * Most of the times
  * I did not receive any notifications
Time Frame: Day 7 +/- 2 days (Visit 2)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers With Single Application of Phenethylamines (D1) | Healthy Volunteers With Single Application of Benzodiazepines (D2) | Healthy Volunteers With Single Application of Cannabinoids (D3) | Healthy Volunteers With Single Application of Opioids (D4)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  Yes | 2 | 4 | 2 | 4
  Most of the times | 2 | 0 | 2 | 0
  I did not receive any notifications | 8 | 8 | 8 | 8

16. Secondary Outcome: Usability Questionnaire - Question 12
Description: User-friendliness of Previct Drugs evaluated by the subject at visit 2. Question 12. Did you notice any issues during usage of Previct Drugs?
  Response options:
  * No
  * Yes
Time Frame: Day 7 +/- 2 days (Visit 2)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers With Single Application of Phenethylamines (D1) | Healthy Volunteers With Single Application of Benzodiazepines (D2) | Healthy Volunteers With Single Application of Cannabinoids (D3) | Healthy Volunteers With Single Application of Opioids (D4)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  No | 5 | 9 | 3 | 8
  Yes | 7 | 3 | 9 | 4

17. Secondary Outcome: Usability Questionnaire - Question 13
Description: User-friendliness of Previct Drugs evaluated by the subject at visit 2. Question 13. Did you require any assistance from the study personnel (e.g., through phone) during the usage of Previct Drugs?
  Response options:
  * Yes
  * No
Time Frame: Day 7 +/- 2 days (Visit 2)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers With Single Application of Phenethylamines (D1) | Healthy Volunteers With Single Application of Benzodiazepines (D2) | Healthy Volunteers With Single Application of Cannabinoids (D3) | Healthy Volunteers With Single Application of Opioids (D4)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  Yes | 0 | 1 | 2 | 2
  No | 12 | 11 | 10 | 10

18. Secondary Outcome: Usability Questionnaire - Question 15
Description: User-friendliness of Previct Drugs evaluated by the subject at visit 2. Question 15. If Yes (to question 13), how often did you require assistance?
  Response options:
  * One occasion
  * Several occasions
  * Most occasions
  * All occasions
Time Frame: Day 7 +/- 2 days (Visit 2)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers With Single Application of Phenethylamines (D1) | Healthy Volunteers With Single Application of Benzodiazepines (D2) | Healthy Volunteers With Single Application of Cannabinoids (D3) | Healthy Volunteers With Single Application of Opioids (D4)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  One occasion | 0 | 0 | 0 | 0
  Several occasions | 0 | 1 | 2 | 2
  Most occasions | 0 | 0 | 0 | 0
  All occasions | 0 | 0 | 0 | 0
  Missing | 1 | 0 | 0 | 0
  Not applicable | 11 | 11 | 10 | 10

19. Secondary Outcome: Usability Questionnaire - Question 16
Description: User-friendliness of Previct Drugs evaluated by the subject at visit 2. Question 16. When starting a measurement, how was your experience finding the right conditions to start the measurement?
  Response options:
  * Very easy
  * Easy
  * Nor easy or difficult
  * Difficult
  * Very difficult
Time Frame: Day 7 +/- 2 days (Visit 2)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers With Single Application of Phenethylamines (D1) | Healthy Volunteers With Single Application of Benzodiazepines (D2) | Healthy Volunteers With Single Application of Cannabinoids (D3) | Healthy Volunteers With Single Application of Opioids (D4)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  Very easy | 1 | 1 | 3 | 2
  Easy | 7 | 10 | 6 | 6
  Nor easy or difficult | 4 | 1 | 3 | 4
  Difficult | 0 | 0 | 0 | 0
  Very difficult | 0 | 0 | 0 | 0

20. Secondary Outcome: Usability Questionnaire - Question 18
Description: User-friendliness of Previct Drugs evaluated by the subject at visit 2. Question 18. How did you experience performing a Nystagmus (look to your extreme right and left) test?
  Response options:
  * Very easy to perform
  * Easy to perform
  * Nor easy or difficult to perform
  * Difficult to perform
  * Very difficult to perform
Time Frame: Day 7 +/- 2 days (Visit 2)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers With Single Application of Phenethylamines (D1) | Healthy Volunteers With Single Application of Benzodiazepines (D2) | Healthy Volunteers With Single Application of Cannabinoids (D3) | Healthy Volunteers With Single Application of Opioids (D4)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  Very easy to perform | 5 | 6 | 6 | 4
  Easy to perform | 6 | 6 | 5 | 6
  Nor easy or difficult to perform | 1 | 0 | 1 | 2
  Difficult to perform | 0 | 0 | 0 | 0
  Very difficult to perform | 0 | 0 | 0 | 0

21. Secondary Outcome: Usability Questionnaire - Question 20
Description: User-friendliness of Previct Drugs evaluated by the subject at visit 2. Question 20. According to you, how many minutes did a Nystagmus test take (from starting test until analyzed)?
  Response options:
  * < 1 minute
  * 1-2 minutes
  * > 3 minutes
Time Frame: Day 7 +/- 2 days (Visit 2)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers With Single Application of Phenethylamines (D1) | Healthy Volunteers With Single Application of Benzodiazepines (D2) | Healthy Volunteers With Single Application of Cannabinoids (D3) | Healthy Volunteers With Single Application of Opioids (D4)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  < 1 minute | 3 | 3 | 2 | 2
  1-2 minutes | 7 | 6 | 6 | 6
  > 3 minutes | 2 | 3 | 4 | 4

22. Secondary Outcome: Usability Questionnaire - Question 21
Description: User-friendliness of Previct Drugs evaluated by the subject at visit 2. Question 21. How often did you have to redo a Nystagmus test?
  Response options:
  * No occasion
  * One occasion
  * Several occasions
  * Most occasions
  * All occasions
Time Frame: Day 7 +/- 2 days (Visit 2)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers With Single Application of Phenethylamines (D1) | Healthy Volunteers With Single Application of Benzodiazepines (D2) | Healthy Volunteers With Single Application of Cannabinoids (D3) | Healthy Volunteers With Single Application of Opioids (D4)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  No occasion | 7 | 8 | 4 | 1
  One occasion | 5 | 2 | 6 | 5
  Several occasions | 0 | 2 | 2 | 6
  Most occasions | 0 | 0 | 0 | 0
  All occasions | 0 | 0 | 0 | 0

23. Secondary Outcome: Usability Questionnaire - Question 23
Description: User-friendliness of Previct Drugs evaluated by the subject at visit 2. Question 23. In general, how easy is it for you to cross your eyes?
  Response options:
  * Very easy
  * Easy
  * Nor easy or difficult
  * Difficult
  * Very difficult
Time Frame: Day 7 +/- 2 days (Visit 2)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers With Single Application of Phenethylamines (D1) | Healthy Volunteers With Single Application of Benzodiazepines (D2) | Healthy Volunteers With Single Application of Cannabinoids (D3) | Healthy Volunteers With Single Application of Opioids (D4)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  Very easy | 5 | 6 | 4 | 4
  Easy | 4 | 3 | 3 | 2
  Nor easy or difficult | 2 | 2 | 3 | 4
  Difficult | 1 | 1 | 2 | 2
  Very difficult | 0 | 0 | 0 | 0

24. Secondary Outcome: Usability Questionnaire - Question 24
Description: User-friendliness of Previct Drugs evaluated by the subject at visit 2. Question 24. How did you experience performing a Cross Eyes test?
  Response options:
  * Very easy to perform
  * Easy to perform
  * Nor easy or difficult to perform
  * Difficult to perform
  * Very difficult to perform
Time Frame: Day 7 +/- 2 days (Visit 2)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers With Single Application of Phenethylamines (D1) | Healthy Volunteers With Single Application of Benzodiazepines (D2) | Healthy Volunteers With Single Application of Cannabinoids (D3) | Healthy Volunteers With Single Application of Opioids (D4)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  Very easy to perform | 5 | 5 | 4 | 5
  Easy to perform | 5 | 6 | 4 | 3
  Nor easy or difficult to perform | 2 | 0 | 2 | 3
  Difficult to perform | 0 | 1 | 2 | 1
  Very difficult to perform | 0 | 0 | 0 | 0

25. Secondary Outcome: Usability Questionnaire - Question 26
Description: User-friendliness of Previct Drugs evaluated by the subject at visit 2. Question 26. According to you, how many minutes did a Cross Eyes test take (from starting until analyzed)?
  Response options:
  * < 1 minute
  * 1-2 minutes
  * > 3 minutes
Time Frame: Day 7 +/- 2 days (Visit 2)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers With Single Application of Phenethylamines (D1) | Healthy Volunteers With Single Application of Benzodiazepines (D2) | Healthy Volunteers With Single Application of Cannabinoids (D3) | Healthy Volunteers With Single Application of Opioids (D4)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  < 1 minute | 4 | 6 | 1 | 4
  1-2 minutes | 7 | 5 | 7 | 7
  > 3 minutes | 1 | 1 | 4 | 1

26. Secondary Outcome: Usability Questionnaire - Question 27
Description: User-friendliness of Previct Drugs evaluated by the subject at visit 2. Question 27. How often did you have to redo a Cross Eyes test?
  Response options:
  * No occasion
  * One occasion
  * Several occasions
  * Most occasions
  * All occasions
Time Frame: Day 7 +/- 2 days (Visit 2)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers With Single Application of Phenethylamines (D1) | Healthy Volunteers With Single Application of Benzodiazepines (D2) | Healthy Volunteers With Single Application of Cannabinoids (D3) | Healthy Volunteers With Single Application of Opioids (D4)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  No occasion | 10 | 9 | 7 | 6
  One occasion | 2 | 2 | 3 | 2
  Several occasions | 0 | 1 | 2 | 4
  Most occasions | 0 | 0 | 0 | 0
  All occasions | 0 | 0 | 0 | 0

27. Secondary Outcome: Usability Questionnaire - Question 29
Description: User-friendliness of Previct Drugs evaluated by the subject at visit 2. Question 29. How did you experience performing a Contraction test?
  Response options:
  * Very easy to perform
  * Easy to perform
  * Nor easy or difficult to perform
  * Difficult to perform
  * Very difficult to perform
Time Frame: Day 7 +/- 2 days (Visit 2)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers With Single Application of Phenethylamines (D1) | Healthy Volunteers With Single Application of Benzodiazepines (D2) | Healthy Volunteers With Single Application of Cannabinoids (D3) | Healthy Volunteers With Single Application of Opioids (D4)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  Very easy to perform | 2 | 2 | 4 | 1
  Easy to perform | 6 | 5 | 5 | 5
  Nor easy or difficult to perform | 4 | 2 | 2 | 5
  Difficult to perform | 0 | 3 | 0 | 0
  Very difficult to perform | 0 | 0 | 1 | 1

28. Secondary Outcome: Usability Questionnaire - Question 31
Description: User-friendliness of Previct Drugs evaluated by the subject at visit 2. Question 31. How was your experience turning your mobile when asked to?
  Response options:
  * Very easy to perform
  * Easy to perform
  * Nor easy or difficult to perform
  * Difficult to perform
  * Very difficult to perform
Time Frame: Day 7 +/- 2 days (Visit 2)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers With Single Application of Phenethylamines (D1) | Healthy Volunteers With Single Application of Benzodiazepines (D2) | Healthy Volunteers With Single Application of Cannabinoids (D3) | Healthy Volunteers With Single Application of Opioids (D4)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  Very easy to perform | 5 | 7 | 6 | 4
  Easy to perform | 5 | 3 | 6 | 6
  Nor easy or difficult to perform | 1 | 2 | 0 | 2
  Difficult to perform | 1 | 0 | 0 | 0
  Very difficult to perform | 0 | 0 | 0 | 0

29. Secondary Outcome: Usability Questionnaire - Question 33
Description: User-friendliness of Previct Drugs evaluated by the subject at visit 2. Question 33. According to you, how many minutes did a Contraction test take (from starting test until analyzed)?
  Response options:
  * < 1 minute
  * 1-2 minutes
  * > 3 minutes
Time Frame: Day 7 +/- 2 days (Visit 2)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers With Single Application of Phenethylamines (D1) | Healthy Volunteers With Single Application of Benzodiazepines (D2) | Healthy Volunteers With Single Application of Cannabinoids (D3) | Healthy Volunteers With Single Application of Opioids (D4)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  < 1 minute | 4 | 0 | 1 | 1
  1-2 minutes | 5 | 9 | 8 | 7
  > 3 minutes | 3 | 3 | 3 | 4

30. Secondary Outcome: Usability Questionnaire - Question 34
Description: User-friendliness of Previct Drugs evaluated by the subject at visit 2. Question 34. How often did you have to redo a Contraction test?
  Response options:
  * No occasion
  * One occasion
  * Several occasions
  * Most occasions
  * All occasions
Time Frame: Day 7 +/- 2 days (Visit 2)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers With Single Application of Phenethylamines (D1) | Healthy Volunteers With Single Application of Benzodiazepines (D2) | Healthy Volunteers With Single Application of Cannabinoids (D3) | Healthy Volunteers With Single Application of Opioids (D4)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  No occasion | 5 | 2 | 5 | 3
  One occasion | 3 | 4 | 6 | 2
  Several occasions | 4 | 4 | 0 | 5
  Most occasions | 0 | 2 | 0 | 1
  All occasions | 0 | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: From signed informed consent to study completion, an average of 10 days.
Groups:
- Healthy Volunteers With Single Application of Benzodiasepines (D2): Evaluation of performance, safety, and usability of Previct Drugs when used in healthy volunteers allocated to one out of four medicinal products at Visit 2 to simulate drug use. Benzodiasepines (D2) allocated to this specific group.
Arm/Group | Healthy Volunteers With Single Application of Phenethylamines (D1) | Healthy Volunteers With Single Application of Benzodiasepines (D2) | Healthy Volunteers With Single Application of Cannabinoids (D3) | Healthy Volunteers With Single Application of Opioids (D4)
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 7/12 | 4/12 | 9/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Volunteers With Single Application of Phenethylamines (D1) (N=12) | Healthy Volunteers With Single Application of Benzodiasepines (D2) (N=12) | Healthy Volunteers With Single Application of Cannabinoids (D3) (N=12) | Healthy Volunteers With Single Application of Opioids (D4) (N=12)
Sleepiness (Investigations) | 1 (1) | 2 (2) | 1 (1) | 5 (5) — Due to drug intake.
Double vision (Eye disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Light headed, dizzy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (5)
Vasovagal reaction (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Nausea (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 6 (6)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/99/NCT05731999/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/99/NCT05731999/SAP_001.pdf